CLINICAL TRIAL: NCT04204447
Title: A Prospective Study Showing the Effect of Video Interactive Education on Medical Decision Making in Patients on Opiate Replacement Therapy (ORT) With a History of Hepatitis C
Brief Title: Hepatitis C-Video vs. Brochure Education Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Andrew Talal, Principal Investigator, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002677
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brochure intervention (Experimental): Subjects will be asked to read an educational brochure about Hepatitis C
  Interventions: Other: Hepatitis C Educational Brochure
- Video intervention (Experimental): Subjects will be asked to watch an educational video about Hepatitis C
  Interventions: Other: Hepatitis C Educational Video

INTERVENTIONS:
Other: Hepatitis C Educational Brochure — Subjects will receive information about Hepatitis C through a brochure
  Arms: Brochure intervention
Other: Hepatitis C Educational Video — Subjects will receive information about Hepatitis C through a video
  Arms: Video intervention

SUMMARY:
The purpose of this study is to determine the most effective way to give patients information regarding hepatitis C virus infection. The investigators plan to compare the information retained by some patients who are given a brochure alone versus patients who watch an interactive video about hepatitis C.

DETAILED DESCRIPTION:
Subjects will complete 3 questionnaires, including one about knowledge of Hepatitis C. The subject will then either watch a video or read a brochure about Hepatitis C, then take the same questionnaire again. The subject will then return in one month to take the Hepatitis C questionnaire again.

ELIGIBILITY:
Inclusion Criteria:

* Currently on active treatment for opioid addiction/use
* English as primary language

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Talal, MD, Principal Investigator — SUNY University at Buffalo
Locations (2):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - BestSelf Behavioral Health, Orchard Park, New York

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Talal AH, Ding YX, Markatou M. Innovations in education: A prospective study of storytelling narratives to enhance hepatitis C virus knowledge among substance users. World J Hepatol. 2022 May 27;14(5):972-983. doi: 10.4254/wjh.v14.i5.972. PMID 35721284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brochure Intervention | Video Intervention
Started | 90 | 86
Completed | 83 | 81
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brochure Intervention | Video Intervention | Total
Number analyzed (Participants) | 90 | 86 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (11) | 41 (12) | 42 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 51 | 106
  Male | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: row population totals when summed do equal overall population
  Participants
    Other race: American Indian or Alaska Native | 1 | 0 | 1
    Other race: Asian | 0 | 0 | 0
    Other race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other race: Black or African American | 12 | 1 | 13
    Other race: White | 76 | 74 | 150
    Other race: More than one race | 0 | 0 | 0
    Other race: Unknown or Not Reported | 1 | 11 | 12

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Scores on HCV Knowledge Questionnaire
Description: The main outcome measure was a change in the mean score on a 25-item HCV knowledge assessment without subscales. The instrument values ranged from 0 to 25 with one point per correct answer to questions directly arising from the information contained in the video. One point was assigned to each correct answer, and an increase in the score indicated more correct responses.
Time Frame: Pre-intervention, Immediate post-intervention, and 1 mo. follow up
Measure: Mean (Standard Deviation); unit: Improvement in scores
Arm/Group | Brochure Intervention | Video Intervention
Number analyzed (Participants) | 90 | 86
Improvement in scores
  Pre-intervention | 18.45 (.3) | 19 (0.25)
  Immiediate post-intervention | 20.3 (.35) | 21.75 (0.3)
  One month post-intervention | 20.2 (.3) | 21.7 (0.2)

ADVERSE EVENTS:
Time Frame: 4-6 weeks-Time between the pre-intervention assessment and the post-intervention assessment obtained one month post-intervention.
Description: There were no adverse events in this study.
Arm/Group | Video Intervention | Brochure Intervention
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/90
Other Adverse Events (participants affected / at risk) | 0/86 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04204447/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04204447/SAP_001.pdf